CLINICAL TRIAL: NCT04290091
Title: Detection of Coronary Artery Disease With Micro Electro-Mechanical Sensors
Acronym: DECADE
Status: Completed | Type: Observational
Sponsor: Precordior Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: DECADE
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with CAD: Patients who have hemodynamically significant CAD.
- Patients without CAD: Patients who don't have hemodynamically significant CAD.

SUMMARY:
This study aims to validate the sensor data of gyroscope and accelerometer in detection of hemodynamically significant CAD.

DETAILED DESCRIPTION:
Heart diseases are the most common cause of morbidity and mortality in the western world. Coronary artery disease (CAD) alone is estimated to affect 110 million people globally and resulted in 8.9 million deaths in 2015.

A hallmark phenomenon in the development of CAD is the formation of arterial stenoses eventually limiting the arterial circulation. Myocardial ischemia caused by the stenoses may present symptoms considered typical, i.e, angina pectoris chest pain, but the symptoms may vary up to an asymptomatic state. Estimating the pre-test likelihood of angiographically significant CAD (≥50% diameter stenotic CAD) is a fundamental component in the initial evaluation of symptomatic patients presenting with suspected CAD. This determination directly influences subsequent decisions for noninvasive diagnostic testing and treatment. However, studies have shown a relatively low prevalence of either ischemia or obstructive CAD on noninvasive imaging and invasive angiography (IA) in this population. Therefore, additional methods are needed to improve patient selection for such testing.

Mechanocardiography (MCG) assesses the condition of the heart by measuring the mechanical activity (cardiac muscle motion) of the heart from the surface of thorax. MCG can be measured with accelerometer and gyroscope which react to recoil and vibration caused my cardiac contraction.

This study aims to validate how the gyroscope and accelerometer derived parameters can identify patients with hemodynamically significant CAD in combined contrast computed tomography (CT) coronary angiography and positron emission tomography (PET) perfusion imaging in combination of high-sensitive troponin testing. The performance of different MCG algorithms will be tested offline as a head-to-head comparison with medical history, cardiovascular events, high-sensitive troponin values, coronary computed tomography angiography (CCTA) and PET scan results.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients visiting hospital for suspected CAD and undergoing CCTA
* Signed informed consent as an acceptance to participate to the trial

Exclusion Criteria:

* informed consent not signed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study includes patients who are referred to a CCTA imaging in Turku University hospital, Turku, Finland due to suspected CAD.
Sampling Method: Non-Probability Sample
Enrollment: 930 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Coronary artery disease | Time of enrolment
  CCTA results with optional myocardial PET perfusion imaging

SECONDARY OUTCOMES:
Coronary artery disease event | 1 year after enrolment to the study
  Registry search of hospitalisation due to cardiovascular events
Coronary artery disease event | 2 year after enrolment to the study
  Registry search of hospitalisation due to cardiovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Juhani Knuuti, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haddad F, Saraste A, Santalahti KM, Pankaala M, Kaisti M, Kandolin R, Simonen P, Nammas W, Jafarian Dehkordi K, Koivisto T, Knuuti J, Mahaffey KW, Blomster JI. Smartphone-Based Recognition of Heart Failure by Means of Microelectromechanical Sensors. JACC Heart Fail. 2024 Jun;12(6):1030-1040. doi: 10.1016/j.jchf.2024.01.022. Epub 2024 Apr 3. PMID 38573263